CLINICAL TRIAL: NCT00361010
Title: A Pilot Study of Efficacy and Tolerability of Levetiracetam Monotherapy in Subjects With Childhood Absence Epilepsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: UCB Pharma (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KeppraCAE
Record Dates: First submitted 2006-08-03; First posted 2006-08-07 (Estimated); Last update posted 2011-07-28 (Estimated); Status verified 2011-07

CONDITIONS: Epilepsy; Childhood Absence Epilepsy; Seizures
Keywords: Keppra; Epilepsy; Childhood Absence Epilepsy; Seizures
MeSH Terms: conditions — Epilepsy; Epilepsy, Absence; Seizures | interventions — Levetiracetam

INTERVENTIONS:
Drug: Levetiracetam

SUMMARY:
Childhood absence epilepsy (CAE) is a form of generalized epilepsy syndrome. Clinically these seizures are manifest with a sudden, brief (3-15 second) loss of awareness followed by a quick recovery to baseline. Keppra (levetiracetam) is approved by the U.S. Food and Drug Administration (FDA) to treat partial seizures in adults. It is currently being studied in children with partial seizures. Absence seizures can be difficult to detect clinically, therefore the response to therapy will be determined both by clinical observation and by 24 hour EEG recordings. The researchers hope that with this information they will learn how well it works for the treatment of childhood absence epilepsy and at what dose. This is an open-label, dose-ranging pilot study of levetiracetam in subjects with newly diagnosed childhood absence epilepsy. Approximately 20 patients will be needed to study effectiveness and dose requirements. Subjects must not be on any antiepileptic medication at the time of entry into the study. Male and female subjects from the ages of 4 to 10 years of age may participate.

DETAILED DESCRIPTION:
This is a 12 week ( 12 week treatment phase), dose ranging pilot study on the effectiveness of levetiracetam for the treatment of childhood absence epilepsy. It consists of 1 phase. The treatment phase where the optimal medication dose will be defined. Absence seizures are often brief and subtle with no postictal manifestations. As a result, clinical observation alone is inadequate to assess the seizure Therefore, both subjective clinical response (parental/caregiver assessment) and EEG recordings are an important part of evaluation of treatment response. A 6 hour outpatient video-EEG study (including 3 minutes of hyperventilation), followed by an 18 hour ambulatory EEG recording - for total 24 hour EEG recording will be done before treatment and every 2 weeks after each dose plateau is reached )

ELIGIBILITY:
Inclusion Criteria:

* CAE by EEG criteria
* Naive to antiepileptics
* Onset 3 to 10 years old
* A history of daily seizures
* Age between 4 and 10
* Weight at least 5th percentile for age
* Be able to take oral medications
* Be willing to return for diagnostic testing and visits and adhere to medication regime

Exclusion Criteria:

* An EEG with any of the following abnormalities
* Focal epilepsy
* Slow spike and wave discharges
* Photoconvulsive response
* Slow background rhythms for age
* Currently being treated with an antiepileptic drug (AED)
* History of MR
* A history of myoclonic, atonic,tonic or astatic seizures
* A clinically unstable disease

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2006-12; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
The primary efficacy variable will be change in seizure frequency.

SECONDARY OUTCOMES:
Determine the design of a larger placebo controlled monotherapy study of the use of levetiracetam for CAE.

CONTACTS AND LOCATIONS:
Overall Officials: Deepak K Lachhwani, MD, Principal Investigator — The Cleveland Clinic, Division of Pediatric Neurology
Locations (2):
- United States (2):
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - The Cleveland Clinic, Cleveland, Ohio